CLINICAL TRIAL: NCT05386056
Title: A Phase II Study to Explore the Efficacy and Safety of Pembrolizumab and Photodynamic Therapy in Metastatic Esophageal Squamous Cell Carcinoma Failed at Least One Line of Systemic Treatment
Brief Title: Pembrolizumab and Photodynamic Therapy in Previously Treated Metastatic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021YJZ100
Record Dates: First submitted 2022-05-11; First posted 2022-05-23 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Pembrolizumab; Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Photodynamic Therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; sinoporphyrin sodium; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Pembrolizumab plus photodynamic therapy (PDT) (Experimental): Interventions:
  * Drug: Pembrolizumab
  * Drug: sinoporphyrin sodium (DVDMS)
  * Photodynamic therapy (PDT)
  Interventions: Drug: Pembrolizumab; Drug: Sinoporphyrin Sodium; Procedure: Photodynamic therapy

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg administered IV Q3W on Day 1 of each 3-week cycle, up to 35 administrations.
  Other Names: MK-3475
Drug: Sinoporphyrin Sodium — 0.2mg/kg, intravenously on day -2 of cycle 1.
  Other Names: DVDMS
Procedure: Photodynamic therapy — PDT to primary site of ESCC will be given on day -1 of the treatment (24 hours after injection of DVDMS).
  Other Names: PDT

SUMMARY:
This is a phase 2 trial investigating the effect and safety of pembrolizumab and photodynamic therapy (PDT) in metastatic esophageal squamous cell carcinoma failed at least one line of systemic treatment.

The primary efficacy hypotheses are that the objective response rate (ORR) of combination of PDT and pembrolizumab could be improved compared with pembrolizumab for both primary and metastatic lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of esophageal squamous cell carcinoma with metastasis/metastases who failed at least one line of systemic treatment for metastatic disease.
2. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
3. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: a. Not a woman of childbearing potential (WOCBP) OR b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Have measurable disease based on RECIST 1.1.
6. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
8. Have adequate organ function.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Include but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV) infection.
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as hepatitis C virus RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a known history of active TB (Bacillus Tuberculosis).
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 in all participants | Up to 2 years
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. For this analysis, ORR will be assessed in all participants who receive at least 1 dose of pembrolizumab.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) per RECIST 1.1 in all participants | Up to 2 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first. For this analysis, PFS will be assessed in all participants who receive at least 1 dose of pembrolizumab.
Overall Survival (OS) in all participants | Up to 2 years
  OS is defined as the time from randomization to death due to any cause. For this analysis, OS will be assessed in all participants who receive at least 1 dose of pembrolizumab.
Incidence of Treatment-Related Adverse Events | Until 30 days after the last treatment
  An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. The number of participants who experienced ≥1 AE will be presented.
Change from baseline in the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30) Score | Baseline, and 6 months
  The EORTC QLQ-C30 was developed to assess the quality of life of patients with cancer. It contains 30 questions (items), 24 of which aggregate into nine multi-item scales representing various aspects, or dimensions, of quality of life (QOL): one global scale, five functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, nausea, pain), and six additional single-symptom items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhoea) and perceived financial impact of the disease. Individual items are scored on a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Raw scores for each scale are standardized into a range of 0 to 100 by linear transformation; a higher score on the global and functional scales represents a higher ("better") level of functioning, and a higher score on the symptom scale represents a higher ("worse") level of symptoms.
Change from baseline in the EORTC Quality Of Life Questionnaire Oesophageal Module (QLQ-OES18) Score | Baseline, and 6 months
  The EORTC QLQ-OES18 is a disease-specific questionnaire developed and validated to address measurements specific to esophageal cancer. It contains 18 items and is based on four subscales-dysphagia (three items), eating (four items), reflux (two items) and pain (three items), as well as six single-item subscales-saliva swallowing, choking, dry mouth, taste, cough and speech. All items are scored using a four-point Likert scale that offers these response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. Raw scores are standardized into a range of 0 to 100 by linear transformation; higher symptom scores represent a higher ("worse") level of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No